CLINICAL TRIAL: NCT02496182
Title: Pirfenidone in the Chronic Hypersensitivity Pneumonitis Treatment
Acronym: Picheon
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Medifarma, S. A. de C. V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C34-11
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Alveolitis Extrinsic Allergic; Pulmonary Fibrosis
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic; Pulmonary Fibrosis | interventions — Excipients; pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Conventional treatment (Prednisone 0.5 mg/kg/day for 4 weeks, then 0.25 mg/Kg/day for 8 weeks and maintenance dosage of 0.125 mg/Kg/day plus Azathioprine 2-3 mg/kg/day with a maximal dosage of 150 mg/day starting with 25-50 mg/day increasing gradually until day 14 with maximal dosage) plus Placebo tablet 2 times at day.
  Interventions: Drug: Placebo
- Pirfenidone 1800 mg (Experimental): Conventional treatment (0.5 mg/kg/day for 4 weeks, then 0.25 mg/Kg/day for 8 weeks and maintenance dosage of 0.125 mg/Kg/day plus Azathioprine 2-3 mg/kg/day with a maximal dosage of 150 mg/day starting with 25-50 mg/day increasing gradually until day 14 with maximal dosage) plus Pirfenidone long release tablet 900 mg 2 times at day, starting with 600 mg at day
  Interventions: Drug: Pirfenidone
- Pirfenidone 1200 mg (Experimental): Conventional treatment (0.5 mg/kg/day for 4 weeks, then 0.25 mg/Kg/day for 8 weeks and maintenance dosage of 0.125 mg/Kg/day plus Azathioprine 2-3 mg/kg/day with a maximal dosage of 150 mg/day starting with 25-50 mg/day increasing gradually until day 14 with maximal dosage) plus Pirfenidone long release tablet 600 mg 2 times at day starting with 600 mg at day
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Placebo — Placebo tablet only with the excipients of the Pirfenidone tablet
  Other Names: Excipient Tablet
  Arms: Placebo
Drug: Pirfenidone — Conventional Treatment (Prednisone+Azathioprine) plus Pirfenidone 1800 mg
  Other Names: Kitoscell LP
  Arms: Pirfenidone 1800 mg
Drug: Pirfenidone — Conventional Treatment (Prednisone+Azathioprine) plus Pirfenidone 1200 mg
  Other Names: KitosCell LP
  Arms: Pirfenidone 1200 mg

SUMMARY:
The Chronic Hypersensitivity Pneumonitis (HP), is an inflammatory disease who has an evolution to develop progressive interstitial fibrosis, who cause the death of the patient. Actually HP has been treated with Prednisone and occasionally with Azathioprine, but unfortunately the treatment with these drugs have not an effective result to treat the interstitial fibrosis.

Pirfenidone has been studied over the world for the treatment of Fibrotic diseases, with positive results, and due to the Pirfenidone mechanism of action has anti-inflammatory and anti-fibrotic properties, the investigators propose to evaluate the addition of Pirfenidone to the actual treatment with Prednisone and Azathioprine in the treatment of patients with Pulmonary Fibrosis secondary to a Chronic Hypersensitivity Pneumonitis.

DETAILED DESCRIPTION:
The Chronic Hypersensitivity Pneumonitis (HP), is a complex syndrome due to a exaggerated immune response caused by inhalation of foreign substances, such as molds, dusts, and organic particles, causing alveoli inflammation and in the chronic forms the disease has high rate of mortality, due to the big number of patients who develop progressive interstitial fibrosis and eventually they curse with respiratory insufficiency who cause the death of the patient.

Pirfenidone has been studied over the world for the treatment of Idiophatic Pulmonary Fibrosis (IPF), disease who constitute the most aggressive of the fibrotic diseases of the lung. Additionally Pirfenidone has been showed potential results in the treatment of fibrotic diseases in other organs, as Liver, Kidney, Hearth, etc. Pirfenidone has been described as a modulator of the fibrotic process due to his action over TGF-beta and MMP´s and also has into-inflammatory actions acting over TNF-alfa and IL-1 and IL-6.

Actually HP has been treated with Prednisone and occasionally with Azathioprine, but a high number of patients will develop irreversibly to a interstitial fibrosis with pulmonary parenchyma destruction. Unfortunately the investigators have not an effective treatment for this cases. Due to the positive results obtained with Pirfenidone in the treatment of IPF and other kind of organ fibrosis, the investigators propose to evaluate the addition of Pirfenidone to the treatment with Prednisone and Azathioprine in the treatment of patients with Pulmonary Fibrosis secondary to a Chronic Hypersensitivity Pneumonitis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hypersensitivity pneumonitis with recent diagnosis confirmed by HRT with or without biopsy
* Acceptation with signed informed consent

Exclusion Criteria:

* No confirmed diagnosis
* Patients with peptic ulcer
* Pregnancy or breast feeding period
* Clinical signs of active infection
* History of severe Hepatic disease
* History of severe Kidney disease, who requires some kind of dialysis
* History of inestable cardiopathy
* History of alcohol or drugs abuse
* Bronchial hyperactivity or History of asthma or EPOC
* Smoking habit 3 months before the starting or patient who decline suspend the smoking habit during the study
* Patient with impossibility to make spirometry or who can not walk
* Use of Immunosuppressants, cytotoxic agents, cytosine modulators or receptor antagonist, fluvoxamine or daily use of sildenafil.
* Patients who not accept sign the informed consent

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 52 weeks
  The measurement of FVC will be at 26 and 52 weeks

SECONDARY OUTCOMES:
High Resolution Tomography | 52 weeks
  Evaluation of the inflammation and fibrosis grade with the Kazerooni scale
6 minutes walk distance test | 52 weeks
  quantification of the walking distance at 6 minutes
San George Qty Score, SOBQ and EQ5D Quality Scores | 52 weeks
  As a composite outcome to evaluate the quality of life
Pulmonary artery systolic pressure with echocardiogram | 52 weeks
  measurement of pressure
Oxygen desaturation in exercise | 52 weeks
  Measurement of Oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Lacasse Y, Selman M, Costabel U, Dalphin JC, Ando M, Morell F, Erkinjuntti-Pekkanen R, Muller N, Colby TV, Schuyler M, Cormier Y; HP Study Group. Clinical diagnosis of hypersensitivity pneumonitis. Am J Respir Crit Care Med. 2003 Oct 15;168(8):952-8. doi: 10.1164/rccm.200301-137OC. Epub 2003 Jul 3. PMID 12842854
- [Background] Selman M. Hypersensitivity pneumonitis: a multifaceted deceiving disorder. Clin Chest Med. 2004 Sep;25(3):531-47, vi. doi: 10.1016/j.ccm.2004.04.001. PMID 15331190
- [Background] Gaxiola M, Buendia-Roldan I, Mejia M, Carrillo G, Estrada A, Navarro MC, Rojas-Serrano J, Selman M. Morphologic diversity of chronic pigeon breeder's disease: clinical features and survival. Respir Med. 2011 Apr;105(4):608-14. doi: 10.1016/j.rmed.2010.11.026. Epub 2010 Dec 16. PMID 21167698
- [Background] Macias-Barragan J, Sandoval-Rodriguez A, Navarro-Partida J, Armendariz-Borunda J. The multifaceted role of pirfenidone and its novel targets. Fibrogenesis Tissue Repair. 2010 Sep 1;3:16. doi: 10.1186/1755-1536-3-16. PMID 20809935
- [Background] Selman M, Pardo A, Richeldi L, Cerri S. Emerging drugs for idiopathic pulmonary fibrosis. Expert Opin Emerg Drugs. 2011 Jun;16(2):341-62. doi: 10.1517/14728214.2011.565049. Epub 2011 Mar 17. PMID 21410428
- [Background] Schaefer CJ, Ruhrmund DW, Pan L, Seiwert SD, Kossen K. Antifibrotic activities of pirfenidone in animal models. Eur Respir Rev. 2011 Jun;20(120):85-97. doi: 10.1183/09059180.00001111. PMID 21632796
- [Derived] Mateos-Toledo H, Mejia-Avila M, Rodriguez-Barreto O, Mejia-Hurtado JG, Rojas-Serrano J, Estrada A, Castillo-Pedroza J, Castillo-Castillo K, Gaxiola M, Buendia-Roldan I, Selman M. An Open-label Study With Pirfenidone on Chronic Hypersensitivity Pneumonitis. Arch Bronconeumol (Engl Ed). 2020 Mar;56(3):163-169. doi: 10.1016/j.arbres.2019.08.019. Epub 2019 Nov 26. English, Spanish. PMID 31784348